CLINICAL TRIAL: NCT04611802
Title: A Phase 3, Randomized, Observer-Blinded, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine (SARS-CoV-2 rS) With Matrix-M1™ Adjuvant in Adult Participants ≥ 18 Years With a Pediatric Expansion in Adolescents (12 to < 18 Years)
Brief Title: A Study to Evaluate the Efficacy, Immune Response, and Safety of a COVID-19 Vaccine in Adults ≥ 18 Years With a Pediatric Expansion in Adolescents (12 to<18 Years) at Risk for SARS-CoV-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV-301
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV Infection; Covid19
Keywords: Coronavirus; Prevent-19; Booster
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Coronavirus Infections | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; Sodium Chloride; Immunization, Secondary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial vaccination) (Experimental): 2 doses of 5 μg SARS-CoV-2 rS + 50 μg Matrix-M1 adjuvant (co-formulated), 1 dose each on Days 0 and 21 in Initial Vaccination Period.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period)
- Placebo (Initial Vaccination) (Placebo Comparator): 2 doses of Placebo (Saline), 1 dose each on Days 0 and 21in Initial Vaccination Period.
  Interventions: Other: Placebo (Initial Vaccination Period)
- SARS-CoV-2 rS/Matrix-M1 Adjuvant (Crossover Vaccination) (Experimental): One dose of 5 μg SARS-CoV-2 rS + 50 μg Matrix-M1 adjuvant (co-formulated) on Day 0 or Day 21 in Crossover Vaccination Period.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Crossover Vaccination period)
- SARS-CoV-2 rS/Matrix-M1 Adjuvant (Booster Vaccination) (Experimental): One dose of 5 μg SARS-CoV-2 rS + 50 μg Matrix-M1 adjuvant (co-formulated) on Day 0 Booster Vaccination Period.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Booster Vaccination)
- SARS-CoV-2 rS/Matrix-M1 Adjuvant (Second Booster) (Experimental): One dose of 5 μg SARS-CoV-2 rS + 50 μg Matrix-M1 adjuvant (co-formulated) on Day 0 Second Booster Vaccination Period.
  Interventions: Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Second Booster Vaccination)
- Placebo (Crossover Vaccination) (Placebo Comparator): One dose of Placebo (Saline) on Day 0 or Day 21 in Crossover Vaccination Period.
  Interventions: Other: Placebo (Crossover Vaccination period)

INTERVENTIONS:
Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial Vaccination Period) — Alternating intramuscular (deltoid) injections of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) on Days 0 and 21 in Initial Vaccination Period.
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Initial vaccination)
Other: Placebo (Initial Vaccination Period) — Alternating intramuscular (deltoid) injections of placebo (0.5 mL) on Days 0 and 21 in Initial Vaccination Period.
  Other Names: Sodium chloride 0.9% (BP, sterile)
  Arms: Placebo (Initial Vaccination)
Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Crossover Vaccination period) — In Crossover Vaccination period, one dose of intramuscular (deltoid) injection of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) on Day 0 or Day 21
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Crossover Vaccination)
Other: Placebo (Crossover Vaccination period) — In Crossover Vaccination period, one dose of intramuscular (deltoid) injection of placebo (0.5 mL) on Day 0 or Day 21
  Other Names: Sodium chloride 0.9% (BP, sterile)
  Arms: Placebo (Crossover Vaccination)
Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Booster Vaccination) — In Booster Vaccination period, one dose of intramuscular (deltoid) injection of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) on Day 0
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Booster Vaccination)
Biological: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Second Booster Vaccination) — In Second Booster Vaccination period, one dose of intramuscular (deltoid) injection of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) on Day 0
  Other Names: NVX-CoV2373
  Arms: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Second Booster)

SUMMARY:
This is a phase 3, randomized, observer-blinded, placebo-controlled study to evaluate the efficacy, safety, and immunogenicity of SARS-CoV-2 rS with Matrix-M1 adjuvant in adult participants and adolescent participants. Additionally providing a Booster Dose to fully vaccinated participants. A substudy is to be conducted at selected sites to evaluate the safety and immunogenicity of a fourth dose (second booster) of NVX-CoV2373 in adults and adolescents, previously fully vaccinated and subsequently boosted with a third dose (first booster)

DETAILED DESCRIPTION:
This is a Phase 3, randomized, observer-blinded, placebo-controlled study to evaluate the efficacy, safety, and immunogenicity of SARS-CoV-2 rS with Matrix-M1 adjuvant in adult participants ≥ 18 years of age (Adult Main Study) and adolescent participants 12 to <18 years (Pediatric Expansion). Additionally, a Booster Amendment will allow for the evaluation of a booster dose of SARS-CoV-2 rS with Matrix-M1 adjuvant in participants who completed the primary series of active vaccine in the Adult Main Study or Pediatric Expansion, as well as in participants who previously completed the primary series of an authorized/approved COVID-19 vaccine. Additionally, a sub-study conducted at specific sites will allow for the evaluation of a second booster dose of SARS-CoV-2 rS with Matrix-M1 adjuvant in participants who completed the primary series of active vaccine in the Adult Main Study and Pediatric Expansion as well as a booster dose in the Booster Amendment of the study.

ELIGIBILITY:
Inclusion Criteria:

Adult Participants :

Each participant in the Adult Main Study and/or the Booster Amendment must meet all of the following criteria to be enrolled in this study:

1. Adults ≥ 18 years of age at screening who, by virtue of age, race, ethnicity or life circumstances, are considered at substantial risk of exposure to and infection with SARS CoV-2.
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [i.e., hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through 3 months after the last vaccination OR agree to consistently use a medically acceptable method of contraception from at least 28 days prior to enrollment and through 3 months after the last vaccination.
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the first vaccination.
5. Agree to not participate in any other SARS-CoV-2 prevention trial during the study follow-up.
6. For the Booster Amendment only, active participants who received a full dose regimen of active vaccine (SARS-CoV-2 rS with Matrix-M1 adjuvant) or any authorized/approved COVID-19 vaccine are eligible for participation. Such participants must demonstrate receipt by producing valid documentation of vaccination at the booster visit.

Pediatric Participants :

Each participant in the Pediatric Expansion and/or the Booster Amendment must meet all of the following criteria to be enrolled in this study:

1. Pediatric participants 12 to < 18 years of age at screening, determined to be healthy or medically stable by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the first vaccination.
2. Participant and parent(s)/caregiver(s) or legally acceptable representative willing and able to give informed consent and assent, as required, prior to study enrollment and to comply with study procedures.
3. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] must agree to be heterosexually inactive from at least 28 days prior to enrollment and through 3 months after the last vaccination OR agree to consistently use a medically acceptable method of contraception from at least 28 days prior to enrollment and through 3 months after the last vaccination.
4. Agree to not participate in another SARS-CoV-2 prevention trial during the study follow-up.
5. For the Booster Amendment only, active participants who received a full dose regimen of active vaccine (SARS-CoV-2 rS with Matrix-M1 adjuvant) or any authorized/approved COVID-19 vaccine are eligible for participation. Such participants must demonstrate receipt by producing valid documentation of vaccination.

Site-Specific Sub Study:

Each participant in the Substudy must meet all of the following criteria to be enrolled in this study:

1. Be an active, enrolled participant in the 2019nCoV-301 study.
2. Adults 18 years of age or older or adolescents 12 to < 18 years of age at initial screening for the parent study.
3. Willing and able to give informed consent prior to substudy enrollment and to comply with extra study procedures.
4. Documented receipt of the 2 doses of the primary series of NVX-CoV2373 and the booster (third dose) of NVX-CoV2373 in the parent protocol. The booster dose must have been administered at least 6 months prior to entering the substudy.
5. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile or postmenopausal) must agree to be heterosexually inactive from at least 28 days prior to entering and through the end of the substudy OR agree to consistently use a medically acceptable method of contraception for the 28 days of follow-up for the substudy.
6. Is medically stable, as determined by the investigator (based on review of health status, vital signs (to include body temperature) and targeted physical examination (if medically indicated by reported symptoms). Vital signs must be within medically acceptable ranges prior to administration of study vaccination.
7. Agree to not participate in any other non-NVX-CoV2373 study during the substudy.

Note: For participants who develop COVID-19, anti-SARS-CoV-2 therapy (approved, authorized or investigational) is permitted.

Exclusion Criteria:

Adult and adolescent participants meeting any of the following criteria will be excluded from the study:

1. Unstable acute or chronic illness. Criteria for unstable medical conditions include:

   1. Substantive changes in chronic prescribed medication (change in class or significant change in dose) in the past 2 months.
   2. Currently undergoing workup of undiagnosed illness that could lead to diagnosis of a new condition.

   Note: Well-controlled human immunodeficiency virus [HIV] with undetectable HIV RNA [< 50 copies/mL] and CD4 count > 200 cells/µL for at least 1 year, documented within the last 6 months, is NOT considered an unstable chronic illness. Participant's or parent's/caregiver's verbal report will suffice as documentation.
2. Participation in research involving an investigational product (drug/biologic/device) administered within 45 days prior to first study vaccination.
3. History of a previous laboratory-confirmed diagnosis of SARS-CoV-2 infection or COVID-19. A previous diagnosis of COVID-19 during participation in this trial is not exclusionary for the Booster Amendment.
4. Received any vaccine within 4 days prior to first study vaccination or planned receipt of any vaccine before Day 49 (i.e., 28 days after second vaccination), except for influenza vaccination, which may be received ≥ 4 days prior to or ≥ 7 days after either study vaccination. Rabies vaccine, at any time it is medically indicated, is not exclusionary. Prior receipt of another approved or authorized COVID-19 vaccine prior to booster injection is not exclusionary in the Booster Amendment. Such participants must provide documentation of vaccine and date(s) of administration.
5. Autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) or therapy that causes clinically significant immunosuppression. NOTE: Stable endocrine disorders (eg, thyroiditis, pancreatitis, including stable diabetes mellitus) are NOT excluded.
6. Chronic administration (defined as > 14 continuous days) of immunosuppressant or systemic glucocorticoids causing clinically significant immunocompromise, within 90 days prior to first study vaccination and/or third (booster) vaccination. NOTE: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 20 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids is permitted. Topical tacrolimus and ocular cyclosporin are permitted.
7. Received immunoglobulin or blood-derived products, within 90 days prior to first study vaccination and/or third (booster) vaccination.
8. Active cancer (malignancy) on chemotherapy that is judged to cause clinically significant immunocompromise within 1 year prior to first study vaccination (with the exception of malignancy cured via excision, at the discretion of the investigator). This criterion is not applicable to participants diagnosed during participation in this trial who accept participation in the Booster Amendment.
9. Any known allergies to products contained in the investigational product.
10. Participants who are breastfeeding, pregnant, or who plan to become pregnant within 3 months following last study vaccination.
11. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results.
12. Study team member or first-degree relative of any study team member (inclusive of Sponsor, and study site personnel involved in the study).
13. Current participation in any other COVID-19 prevention clinical trial.
14. Adult participants who have not received a full dose of any authorized/approved COVID-19 vaccine and are unable to provide valid documentation of vaccination will be excluded from the Booster Amendment.

Adult and adolescent participants meeting any of the following criteria will be excluded from the substudy:

1. History of laboratory-confirmed (by PCR or other antigen testing) COVID-19 infection ≤ 4 months prior to entering the substudy.
2. Known to be clinically significantly immunocompromised.
3. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to entering substudy.
4. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the end of substudy.
5. History of confirmed myocarditis and/or pericarditis since enrollment to the parent study.
6. Any condition that, in the opinion of the investigator, might pose a health risk to the participant, interfere with protocol compliance or interfere with evaluation of the trial vaccine.
7. Study team member or immediate family member of any study team member (inclusive of Sponsor, CRO, and study site personnel involved in the conduct or planning of the substudy).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33000 (Actual)
Dates: Start 2020-12-27 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Adult Main Study and Pediatric Expansion: Participants with Symptomatic Mild, Moderate, or Severe Coronavirus Disease 2019 (COVID-19) | Day 28 to Day 750
  Number of participants with first occurrence of positive (+) polymerase chain reaction (PCR)-confirmed SARS-CoV-2 illness with symptomatic mild, moderate, or severe COVID-19, with each symptom lasting for at least 2 consecutive days, with onset from Day 28 (7 days after second vaccination dose) through the length of the study.
Pediatric Expansion: Reactogenicity Incidence and Severity | Day 0 to Day 27
  Reactogenicity incidence and severity (mild, moderate or severe) recorded by all participants on their electronic patient-reported outcome diary application (eDiary) on days of vaccination and subsequent 6 days (total 7 days after each vaccine injection).
Pediatric Expansion: Incidence and Severity of Medically Attended Adverse Events (MAAEs) Through Day 49 | Day 0 to Day 49
  Number of participants with mild, moderate, or severe MAAEs through Day 49 i.e. 28 days after second injection of each set of vaccinations (initial and crossover).
Pediatric Expansion: Incidence and Severity of Unsolicited Adverse Events (AEs) Through Day 49 | Day 0 to Day 49
  Number of participants with mild, moderate, or severe AEs through Day 49 i.e. 28 days after second injection of each set of vaccinations (initial and crossover).
Pediatric Expansion: Incidence and Severity of MAAEs Attributed to Study Vaccine Through Specified Time Points | Day 90 to Day 750
  Number of participants with mild, moderate, or severe MAAEs attributed to study vaccine through specified time points approximately every 3 and 6 months.
Pediatric Expansion: Incidence and Severity of Serious Adverse Events (SAEs) Through Specified Time Points | Day 90 to Day 750
  Number of participants with mild, moderate, or severe SAEs attributed to study vaccine through specified time points approximately every 3 and 6 months.
Pediatric Expansion: Incidence and Severity of Adverse Events of Special Interest (AESIs) Through Specified Time Points | Day 90 to Day 750
  Number of participants with mild, moderate, or severe AESIs attributed to study vaccine through specified time points approximately every 3 and 6 months.
Pediatric Expansion: Incidence and Severity of SAEs Attributed to Study Vaccine Through Specified Time Points until Month 24 | Day 90 to Day 750
  Number of participants with mild, moderate, or severe SAEs attributed to study vaccine and AESIs through specified time points until Month 24 or the EoS.
Pediatric Expansion: Incidence and Severity of MAAEs Attributed to Study Vaccine Through Specified Time Points until Month 24 | Day 90 to Day 750
  Number of participants with mild, moderate, or severe MAAEs attributed to study vaccine and AESIs through specified time points until Month 24 or the EoS.
Pediatric Expansion: Incidence and Severity of AESIs Attributed to Study Vaccine Through Specified Time Points until Month 24 | Day 90 to Day 750
  Number of participants with mild, moderate, or severe AESIs attributed to study vaccine and AESIs through specified time points until Month 24 or the EoS.
Pediatric Expansion: Antibodies to SARS-CoV-2 Nucleoprotein (NP) at Specified Time Points | Day 35
  Number of participants with antibodies to SARS-CoV-2 NP at Day 35 to determine natural infection and to determine the incidence of asymptomatic infection acquired during study follow-up.
Pediatric Expansion: Deaths Due to Any Cause | Day 0 to Day 750
  Number of participants who died during the study due to any cause.

SECONDARY OUTCOMES:
Adult Main Study and Pediatric Expansion: Participants with Symptomatic Moderate or Severe COVID-19 | Day 28 to Day 750
  Number of participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness with symptomatic moderate or severe COVID-19, with each symptom lasting for at least 2 consecutive days, with onset from Day 28 (7 days after second vaccination dose) through the length of the study.
Adult Main Study and Pediatric Expansion: Participants with Any Symptomatic COVID-19 | Day 28 to Day 750
  Number of participants with first occurrence of (+) PCR-confirmed SARS-CoV-2 illness with any symptomatic COVID-19, with each symptom lasting for at least 2 consecutive days, with onset from Day 28 (7 days after second vaccination dose) through the length of the study.
Adult Main Study and Pediatric Expansion: Neutralizing Antibody Activity Expressed as Geometric Mean Titers (GMTs) | Day 0 to Day 750
  Neutralizing antibody activity as detected by microneutralization assay (MN) as expressed as GMTs at Days 0, 35 and at specified time points through EoS.
Adult Main Study and Pediatric Expansion: Neutralizing Antibody Activity Expressed as Geometric Mean Fold Rises (GMFRs) | Day 0 to Day 750
  Neutralizing antibody activity as detected by MN as expressed as GMFRs at Days 0, 35 and at specified time points through EoS.
Adult Main Study and Pediatric Expansion: Serum Immunoglobulin G (IgG) Antibody Levels Expressed as GMTs | Day 0 to Day 750
  Serum IgG antibody levels specific to SARS-CoV-2 rS protein antigen(s) as detected by enzyme-linked immunosorbent assay (ELISA) expressed as GMTs at Days 0, 35 and at specified time points through EoS.
Adult Main Study and Pediatric Expansion: Serum IgG Antibody Levels Expressed as GMFRs | Day 0 to Day 750
  Serum IgG antibody levels specific to SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at Days 0, 35 and at specified time points through EoS.
Adult Main Study and Pediatric Expansion: Human Angiotensin-Converting Enzyme 2 (hACE2) Receptor Binding Inhibition Assay Expressed as GMTs | Day 0 to Day 750
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by hACE2 receptor binding inhibition assay expressed as GMTs at Days 0, 35 and at specified time points through EoS.
Adult Main Study and Pediatric Expansion: hACE2 Receptor Binding Inhibition Assay Expressed as GMFRs | Day 0 to Day 750
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by hACE2 receptor binding inhibition assay expressed as GMFRs at Days 0, 35 and at specified time points through EoS.
Adult Main Study and Pediatric Expansion: Serum Immunoglobulin G (IgG) Antibody Levels Expressed as GMTs at Later Time Points | Day 165 to Day 750
  Serum IgG antibody levels specific to SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMTs at Months 6, 12, 18, and 24.
Adult Main Study and Pediatric Expansion: Serum Immunoglobulin G (IgG) Antibody Levels Expressed as GMFRs at Later Time Points | Day 165 to Day 750
  Serum IgG antibody levels specific to SARS-CoV-2 rS protein antigen(s) as detected by ELISA expressed as GMFRs at Months 6, 12, 18, and 24.
Adult Main Study and Pediatric Expansion: hACE2 Receptor Binding Inhibition Assay Expressed as GMTs at Later Time Points | Day 165 to Day 750
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by hACE2 receptor binding inhibition assay expressed as GMTs at Months 6, 12, 18, and 24.
Adult Main Study and Pediatric Expansion: hACE2 Receptor Binding Inhibition Assay Expressed as GMFRs at Later Time Points | Day 165 to Day 750
  Epitope-specific immune responses to the SARS-CoV-2 rS protein receptor binding as detected by hACE2 receptor binding inhibition assay expressed as GMFRs at Months 6, 12, 18, and 24.
Adult Main Study and Pediatric Expansion: Neutralizing Antibody Activity Expressed as GMTs at Later Time Points | Day 165 to Day 750
  Neutralizing antibody activity as detected by MN as expressed as GMTs at Months 6, 12, 18, and 24.
Adult Main Study and Pediatric Expansion: Neutralizing Antibody Activity Expressed as GMFRs at Later Time Points | Day 165 to Day 750
  Neutralizing antibody activity as detected by MN as expressed as GMFRs at Months 6, 12, 18, and 24.
Adult Main Study and Pediatric Expansion: Description of Course, Treatment and Severity of COVID-19 | Day 28 to Day 750
  Description of course, treatment and severity of COVID-19 reported after a PCR-confirmed case via the Endpoint Form.
Adult Main Study: Reactogenicity Incidence and Severity | Day 0 to Day 27
  Reactogenicity incidence and severity (mild, moderate or severe) recorded by all participants on their electronic patient-reported outcome diary application (eDiary) on days of vaccination and subsequent 6 days (total 7 days after each vaccine injection).
Adult Main Study: Incidence and Severity of Medically Attended Adverse Events (MAAEs) Through Day 49 | Day 0 to Day 49
  Number of participants with mild, moderate, or severe MAAEs through Day 49 i.e. 28 days after second injection of each set of vaccinations (initial and crossover).
Adult Main Study: Incidence and Severity of Unsolicited Adverse Events (AEs) Through Day 49 | Day 0 to Day 49
  Number of participants with mild, moderate, or severe AEs through Day 49 i.e. 28 days after second injection of each set of vaccinations (initial and crossover).
Adult Main Study: Incidence and Severity of MAAEs Attributed to Study Vaccine Through Specified Time Points | Day 90 to Day 750
  Number of participants with mild, moderate, or severe MAAEs attributed to study vaccine through specified time points approximately every 3 months.
Adult Main Study: Incidence and Severity of Serious Adverse Events (SAEs) Attributed to Study Vaccine Through Specified Time Points | Day 90 to Day 750
  Number of participants with mild, moderate, or severe SAEs attributed to study vaccine through specified time points approximately every 3 months.
Adult Main Study: Incidence and Severity of Adverse Events of Special Interest (AESIs) Attributed to Study Vaccine Through Specified Time Points | Day 90 to Day 750
  Number of participants with mild, moderate, or severe AESIs attributed to study vaccine through specified time points approximately every 3 months.
Adult Main Study: Incidence and Severity of SAEs Attributed to Study Vaccine Through Specified Time Points until Month 24 | Day 90 to Day 750
  Number of participants with mild, moderate, or severe SAEs attributed to study vaccine and AESIs through specified time points until Month 24 or the EoS.
Adult Main Study: Incidence and Severity of MAAEs Attributed to Study Vaccine Through Specified Time Points until Month 24 | Day 360 to Day 750
  Number of participants with mild, moderate, or severe MAAEs attributed to study vaccine and AESIs through specified time points until Month 24 or the EoS.
Adult Main Study: Incidence and Severity of AESIs Attributed to Study Vaccine Through Specified Time Points until Month 24 | Day 360 to Day 750
  Number of participants with mild, moderate, or severe AESIs attributed to study vaccine and AESIs through specified time points until Month 24 or the EoS.
Adult Main Study and Pediatric Expansion: Antibodies to SARS-CoV-2 Nucleoprotein (NP) at Specified Time Points | Day 0 to Day 750
  Number of participants with antibodies to SARS-CoV-2 NP at Days 0 and 35, or at specified time points through EoS to determine natural infection and to determine the incidence of asymptomatic infection acquired during study follow-up.
Adult Main Study and Pediatric Expansion: Antibodies to SARS-CoV-2 Nucleoprotein (NP) at Any Time Point | Day 0 to Day 750
  Number of participants with antibodies to SARS-CoV-2 NP, regardless of whether the infection was symptomatic.
Adult Main Study: IgG antibodies to SARS-CoV-2 rS at Day 35 After First Crossover Vaccination | Day 35 after the first crossover vaccination
  The ratio of geometric mean IgG antibody concentrations will be computed at Day 35 for the new manufacturing process versus the old manufacturing process using the data collected from 300 active vaccine recipients 18 to ≤ 64 years of age enrolled at selected study sites.
Adult Main Study : Deaths Due to Any Cause | Day 0 to Day 750
  Number of participants who died during the study due to any cause.
Adult Main Study and Pediatric Expansion: Participants with 1st episode of positive Polymerase Chain Reaction (PCR) for Coronavirus Disease 2019 (COVID-19) due to a variant not considered as a "variant of concern/interest" | Day 28 to Day 750
  Number of participants with first episode of PCR-positive COVID-19, as defined under the primary endpoint, shown by gene sequencing to represent a variant not considered as a "variant of concern/interest" according to the CDC Variants Classification.

OTHER OUTCOMES:
Booster Amendment: Participants with symptomatic mild, moderate or severe COVID-19 | Day 0 to Day 7
  First episode of PCR-positive mild, moderate, or severe COVID-19 occurring ≥ 7 days after the third (booster) vaccine dose.
Booster Amendment: Participants with PCR positive moderate-to-severe COVID-19 | Day 0 to Day 7
  First episode of PCR-positive moderate-to-severe COVID-19 occurring ≥ 7 days after the third (booster) vaccine dose.
Booster Amendment: Participants with PCR positive COVID-19 due to a variant not considered "variant of interest/concern" | Day 0 to Day 7
  First episode of PCR-positive COVID-19 occurring ≥7 days after the third (booster) vaccine dose and shown by gene sequencing to represent a variant not considered as a "variant of concern/interest" according to the CDC Variants Classification
Booster Amendment: Participants with PCR positive COVID-19 due to a 'variant of concern/interest" | Day 0 to Day 7
  First episode of PCR-positive COVID-19 occurring ≥7 days after the third (booster) vaccine dose, and shown by gene sequencing to represent a "variant of concern/interest" according to the CDC Variants Classification.
Booster Amendment: Neutralizing antibody activity expressed as GMT | Day 0 to Day 28
  Neutralizing antibody titers from Immunogenicity Population immediately prior and at 28 days after administration of the third (booster) vaccine dose expressed as GMT.
Booster Amendment: Neutralizing antibody activity expressed as GMFR | Day 0 to Day 28
  Neutralizing antibody titers from Immunogenicity Population immediately prior and at 28 days after administration of the third (booster) vaccine dose expressed as GMFR.
Booster Amendment: Serum IgG antibody levels expressed as GMT | Day 0 to Day 28
  Serum levels of IgG to SARS-CoV-2 S protein from Immunogenicity Population immediately prior and at 28 days after administration of the third (booster) vaccine dose expressed as GMT.
Booster Amendment: Serum IgG antibody levels expressed as GMFR | Day 0 to Day 28
  Serum levels of IgG to SARS-CoV-2 S protein from Immunogenicity Population immediately prior and at 28 days after administration of the third (booster) vaccine dose expressed as GMFR.
Booster Amendment: hACE2 receptor binding inhibition assay expressed as GMT | Day 0 to Day 28
  hACE2 inhibition titers from Immunogenicity Population immediately prior and at 28 days after administration of the third (booster) vaccine dose expressed as GMT.
Booster Amendment: hACE2 receptor binding inhibition assay expressed as GMFR | Day 0 to Day 28
  hACE2 inhibition titers from Immunogenicity Population immediately prior and at 28 days after administration of the third (booster) vaccine dose expressed as GMFR.
Booster Amendment: Incidence and severity of unsolicited AE's | Day 0 to Day 28
  Incidence and severity of unsolicited AEs through 28 days after the third (booster) vaccine dose.
Booster Amendment: Incidence and severity of MAAE's, SAE's and AESI's | Day 0 to Day 720
  Incidence and severity of MAAEs attributed to study vaccine, SAEs and AESIs through EoS.
Booster Amendment: Description of course, treatment and severity of COVID-19 | Day 0 to Day 7
  Description of course, treatment and severity of COVID-19 reported after a PCR-confirmed case occurring ≥7 days after the third (booster) vaccine dose via the Endpoint Form.
Booster Amendment: Reactogenicity Incidence and Severity | Day0 to Day 7
  Reactogenicity incidence and severity (mild, moderate or severe) recorded by all participants on their electronic patient-reported outcome diary application (eDiary) on days of the third (booster) vaccination and subsequent 6 days.
Booster Amendment: Deaths Due to Any Cause | Day 0 to Day 720
  Number of participants who died during the study due to any cause.
Site Specific Sub Study: Serum IgG to the SARS-CoV-2 spike protein expressed as GMEU | Day 28
  IgG geometric mean ELISA unit concentrations (EU/ml) to the SARS-CoV-2 spike protein at Day 28 following the second booster dose.
Site Specific Sub Study: Serum IgG antibody expressed as GMFR | Day 28
  IgG Geometric Mean Fold Rises (GMFR) at Day 28 post second booster dose relative to Day 28 post-first booster dose.
Site Specific Sub Study: Serum IgG to the SARS-CoV-2 spike protein expressed as SPR | Day 28
  Proportion of participants who achieve seroresponse (≥ 4-fold increase from pre-second booster baseline) in IgG ELISA unit concentrations to the SARS-CoV-2 spike protein at Day 28 post second booster dose.
Site Specific Sub Study: hACE2 Receptor Binding Inhibition Assay Expressed as GMTs | Day 28
  hACE2 inhibition assay titers (GMTs) at Day 28 post second booster dose.
Site Specific Sub Study: hACE2 Receptor Binding Inhibition Assay Expressed as GMFR | Day 28
  hACE2 GMFR at Day 28 post second booster dose relative to Day 28 post-first booster dose.
Site Specific Sub Study: hACE2 Receptor Binding Inhibition Assay Expressed as SPR | Day 28
  Proportion of participants who achieve seroresponse (≥ 4-fold increase from pre-second booster baseline) in hACE2 inhibition assay titers at Day 28 post-second booster dose.Incidence, severity, and duration of solicited adverse events for the 7 days period following the second booster dose.
Site Specific Sub Study: Microneutralization assay (MN) titers to the SARS-CoV-2 wild type virus expressed as GMTs | Day 28
  MN50 geometric mean titers to the SARS-CoV-2 wild-type virus at Day 28 post second booster dose.
Site Specific Sub Study: Microneutralization assay (MN) titers to the SARS-CoV-2 wild type virus expressed as GMFR | Day 28
  MN50 GMFR at Day 28 post second booster dose relative to Day 28 post-first booster dose.
Site Specific Sub Study: Microneutralization assay (MN) titers to the SARS-CoV-2 wild type virus expressed as SPR | Day 28
  Proportion of participants who achieve seroresponse (≥ 4-fold increase from pre-second booster baseline) in MN50 titers concentrations to the wild-type virus at Day 28 post second booster dose.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (152):
- United States (142):
  - Alabama Clinical Therapeutics, Llc (Pediatric Site), Birmingham, Alabama
  - Accel Research Sites (Adult Site), Birmingham, Alabama
  - Central Research Associates, Inc (Pediatric Site), Birmingham, Alabama
  - The Pain Center of Arizona (Adult Site), Phoenix, Arizona
  - Foothills Research Center-CCT Research (Pediatric Site), Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC (Adult Site), Tempe, Arizona
  - Lynn Institute of the Ozarks (Adult Site), Little Rock, Arkansas
  - Preferred Research Partners, Inc. (Adult Site), Little Rock, Arkansas
  - Anaheim Clinical Trials (Adult Site), Anaheim, California
  - Advanced Clinical Research - Rancho Paseo (Pediatric & Adult Site), Banning, California
  - Coast Clinical Research, LLC (Pediatric Site), Bellflower, California
  - Velocity Clinical Research (Pediatric & Adult Site), Chula Vista, California
  - Premier Health Research Center, Llc (Pediatric Site), Downey, California
  - eStudySite - Corporate Offices (Adult Site), La Mesa, California
  - Paradigm Clinical Research Centers, Inc (Pediatric Site), La Mesa, California
  - WR-PRI, LLC (Adult Site), Los Alamitos, California
  - National Research Institute (Pediatric & Adult Site), Los Angeles, California
  - Orange County Research Institute (Pediatric Site), Ontario, California
  - Empire Clinical Research (Pediatric & Adult Site), Pomona, California
  - University of California Davis Health (Pediatric & Adult Site), Sacramento, California
  - Benchmark Research (Pediatric & Adult Site), Sacramento, California
  - California Research Foundation (Pediatric & Adult Site), San Diego, California
  - Synexus Clinical Research US, Inc. (Adult Site), Vista, California
  - Dignity Health Medical Foundation - Woodland (Adult Site), Woodland, California
  - University of Colorado Clinical and Translational Research Centers (Pediatric & Adult Site), Aurora, Colorado
  - Lynn Institute of the Rockies (Adult Site), Colorado Springs, Colorado
  - Meridian Clinical Research (Pediatric Site), Washington D.C., District of Columbia
  - Howard University Hospital Howard/ University College of Medicine (Adult Site), Washington D.C., District of Columbia
  - University Clinical Research-Deland, LLC dba Accel Research Sites (Pediatric & Adult Site), DeLand, Florida
  - SIMED Health, LLC / SIMED Research (Adult Site), Gainesville, Florida
  - M D Clinical (Adult Site), Hallandale, Florida
  - Jacksonville Center for Clinical Research (Pediatric & Adult Site), Jacksonville, Florida
  - Meridien Research/Accel Research (Pediatric & Adult site), Lakeland, Florida
  - Miami Veterans Affairs Medical Center (Adult Site), Miami, Florida
  - Suncoast Research Associates, LLC (Adult Site), Miami, Florida
  - Acevedo Clinical Research Associates (Pediatric Site), Miami, Florida
  - Clinical Neuroscience Solutions Inc (Pediatric & Adult Site), Orlando, Florida
  - Headlands Research Orlando (Adult Site), Orlando, Florida
  - Synexus Clinical Research US, Inc (Adult Site), Pinellas Park, Florida
  - Asclepes Research Centers (Adult & Pediatric Site), Spring Hill, Florida
  - Tampa Heart & Cardiovascular Center (Adult Site), Tampa, Florida
  - Office Of John S. Curran MD (Adult Site), Tampa, Florida
  - Synexus Clinical Research US, Inc. (Adult Site), The Villages, Florida
  - Comprehensive Clinical Trials, Llc (Pediatric & Adult site), West Palm Beach, Florida
  - Emory University Hospital (Adult Site), Atlanta, Georgia
  - Atlanta - Morehouse School of Medicine (Adult Site), Atlanta, Georgia
  - Synexus Clinical Research US, Inc. (Adult Site), Atlanta, Georgia
  - Atlanta Center for Medical Research (Adult Site), Atlanta, Georgia
  - Tekton Research, Inc. (Pediatric Site), Chamblee, Georgia
  - Columbus Regional Research Institute (Adult Site), Columbus, Georgia
  - Clinical Research Atlanta (Adult Site), Stockbridge, Georgia
  - Advanced Clinical Research (Pediatric & Adult Site), Meridian, Idaho
  - Synexus Clinical Research US, Inc (Adult Site), Chicago, Illinois
  - Cedar Crosse Research Center (Adult Site), Chicago, Illinois
  - Providea Health Partners LLC (Adult Site), Evergreen Park, Illinois
  - Synexus USA (Adult Site), Evansville, Indiana
  - Buynak Clinical Research, P.C. (Pediatric & Adult Site), Valparaiso, Indiana
  - The University of Iowa Hospitals & Clinics (Adult Site), Iowa City, Iowa
  - Meridian Clinical Research (Adult Site), Sioux City, Iowa
  - Johnson County Clin-Trials, Inc. (Pediatric & Adult Site), Lenexa, Kansas
  - Alliance for Multispecialty Research (AMR) (Pediatric Site), Newton, Kansas
  - AMR Wichita East (Formerly Heartland Research Associates) (Pediatric SIte), Wichita, Kansas
  - Kentucky Pediatric/Adult Research (Pediatric Site), Bardstown, Kentucky
  - Brownsboro Park Pediatrics (Pediatric Site), Louisville, Kentucky
  - Meridian Clinical Research Baton Rouge (Pediatric Site), Baton Rouge, Louisiana
  - Meridian Clinical Research, LLC (Adult Site), Baton Rouge, Louisiana
  - Med Pharmics, LLC (Pediatric & Adult Site), Metairie, Louisiana
  - Willis-Knighton Physician Network (Adult Site), Shreveport, Louisiana
  - c/o The Pediatric Center of Frederick LLC (Adult & Pediatric Site), Baltimore, Maryland
  - Beth Israel Deaconess Medical Center (Adult Site), Boston, Massachusetts
  - VA Ann Arbor Healthcare System (Adult Site), Ann Arbor, Michigan
  - Wayne State University/ Children's Hospital of Michigan (Adult Site), Detroit, Michigan
  - University of Minnesota (Adult Site), Minneapolis, Minnesota
  - Synexus Clinical Research US, Inc. (Adult Site), Richfield, Minnesota
  - MedPharmics, LLC-Biloxi (Pediatric & Adult Site), Gulfport, Mississippi
  - The Curators of University of Missouri (Adult Site), Columbia, Missouri
  - Sundance Clinical Research, LLC (Pediatric & Adult Site), St Louis, Missouri
  - Meridian Clinical Research (Adult & Pediatric Site), Norfolk, Nebraska
  - Meridian Clinical Research Associates, LLC (Pediatric & Adult Site), Omaha, Nebraska
  - University Of Nebraska Medical Center (Pediatric & Adult Site), Omaha, Nebraska
  - Synexus Clinical Research US, Inc. (Adult Site), Henderson, Nevada
  - Clinical Research Center of Nevada (Pediatric Site), Las Vegas, Nevada
  - Clinical Research Consortium (Adult Site), Las Vegas, Nevada
  - Meridian Clinical Research (Pediatric Site), Binghamton, New York
  - Stony Brook Responder Vaccine Program (Adult Site), Commack, New York
  - Weill Cornell Chelsea CRS (Adult Site), New York, New York
  - Rochester Clinical Research (Pediatric & Adult Site), Rochester, New York
  - NC TraCS Institute - CTRC; University of North Carolina at Chapel Hill (Pediatric & Adult Site), Chapel Hill, North Carolina
  - The Charlotte-Mecklenburg Hospital Authority d/b/a Atrium Health (Pediatric & Adult Site), Charlotte, North Carolina
  - M3-Emerging Medical Research, LLC (Pediatric & Adult Site), Durham, North Carolina
  - Carolina Institute for Clinical Research (Adult Site), Fayetteville, North Carolina
  - Womack Army Medical Center (Adult Site), Fort Bragg, North Carolina
  - M3 Wake Research, Inc (Adult Site), Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC (Adult Site), Rocky Mount, North Carolina
  - Wake Forest Health Network - Pediatrics - Ford, Simpson, Lively & Rice (Pediatric Site), Salem, North Carolina
  - PMG Research of Wilmington, LLC (Adult Site), Wilmington, North Carolina
  - Synexus Clinical Research, US, Inc. (Adult Site), Akron, Ohio
  - Sterling Research Group, Ltd. (Adult Site), Cincinnati, Ohio
  - Synexus Clinical Research US, Inc. (Adult Site), Cincinnati, Ohio
  - Sterling Research Group, Ltd (Pediatric & Adult Site), Cincinnati, Ohio
  - Dr. Shelly David Senders MD Inc. dba Senders Pediatrics (Pediatric Site), Cleveland, Ohio
  - Velocity Clinical Research (Pediatric & Adult Site), Cleveland, Ohio
  - Aventiv Research Inc (Pediatric Site), Columbus, Ohio
  - Medical Research International (Adult Site), Oklahoma City, Oklahoma
  - Lynn Health Science Institute (Pediatric & Adult Site), Oklahoma City, Oklahoma
  - Velocity Clinical Research (Pediatric & Adult Site), Medford, Oregon
  - Preferred Primary Care Physicians, Inc. (Pediatric Site), Pittsburgh, Pennsylvania
  - The Miriam Hospital (TMH) (Adult Site), Providence, Rhode Island
  - Omega Medical Research, Providence (Pediatric & Adult Site), Warwick, Rhode Island
  - Synexus Clinical Research US, Inc. (Adult Site), Anderson, South Carolina
  - Medical University of South Carolina, SCTR Research Nexus (Adult Site), Charleston, South Carolina
  - Coastal Carolina Research Center (Pediatric Site), North Charleston, South Carolina
  - Spartanburg Medical Research (Pediatric Site), Spartanburg, South Carolina
  - American Indian Clinical Trials Research Network (Pediatric & Adult Site), Eagle Butte, South Dakota
  - Accellacare of Bristol (Pediatric & Adult Site), Bristol, Tennessee
  - WR Clinsearch, LLC (Pediatric & Adult Site), Chattanooga, Tennessee
  - Holston Medical Group (Pediatric Site), Kingsport, Tennessee
  - Accellacare US Inc., d/b/a Accellacare of Knoxville (Adult Site), Knoxville, Tennessee
  - Clinical Neurosciecne Solutions, Inc. dba CNS Healthcare (Pediatric & Adult Site), Memphis, Tennessee
  - Clinical Research Associates (Pediatric Site), Nashville, Tennessee
  - Clinical and Translational Research Center at Meharry Medical College (Adult Site), Nashville, Tennessee
  - Benchmark Research (Pediatric & Adult Site), Austin, Texas
  - Ventavia Research Group, LLC (Pediatric Site), Fort Worth, Texas
  - Benchmark Research (Pediatric & Adult Site), Fort Worth, Texas
  - Ventavia Research Group, LLC (Pediatric Site), Houston, Texas
  - Baylor College of Medicine (Adult Site), Houston, Texas
  - DM Clinical Research - Pediatric Healthcare of NW Houston, P.A. (Pediatric Site), Houston, Texas
  - Texas Center for Drug Development, Inc (Pediatric & Adult Site), Houston, Texas
  - The University Of Texas Medical Branch (Utmb) (Pediatric Site), League City, Texas
  - Centex Studies, Inc (Adult Site), McAllen, Texas
  - Research Your Health (Pediatric & Adult site), Plano, Texas
  - AES San Antonio (Adult Site), San Antonio, Texas
  - University of Texas Health Science Center San Antonio (Adult Site), San Antonio, Texas
  - Tekton Research, Inc. (Pediatric Site), San Antonio, Texas
  - DM Clinical Research (Pediatric & Adult Site), Tomball, Texas
  - Wee Care Pediatrics (Pediatric Site), Layton, Utah
  - Wee Care Pediatrics (Pediatric Site), Syracuse, Utah
  - Advanced Clinical Research (Adult Site), West Jordan, Utah
  - Pediatric Research of Charlottesville, LLC (Pediatric Site), Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc (Pediatric & Adult Site), Newport News, Virginia
  - MultiCare Institute for Research & Innovation (Adult Site), Cheney, Washington
  - University of Washington VTEU (Adult Site), Seattle, Washington
- Mexico (8):
  - PanAmerican Clinical Research Mexico S.A de C.V (Adult Site), Guadalajara, Jalisco
  - Instituto Nacional de Salud Publica (INSP) - Cuernavaca - Centro de Investigacion en Salud Poblacional (CISP) (Adult Site), Cuernavaca, Morelos
  - PanAmerican Clinical Research Mexico (Adult Site), Juriquilla, Querétaro
  - Unidad de Atencion Medica e Investigacion en Salud (UNAMIS) (Adult Site), Mérida, Yucatán
  - CAIMED Investigacion en Salud S.A de C.V (Adult Site), Mexico City
  - Caimed Investigacion en Salud S.A. de C.V. (Adult Site), Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Adult Site), Mexico City
  - FAICIC S. DE R.L. DE C.V. (Adult Site), Veracruz
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc. / CAIMED Cneter (Pediatric & Adult Site), Ponce
  - University of Puerto Rico Medical Sciences Campus Maternal Infant Studies Center (Adult Site), San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deming ME, Brown ER, McArthur MA, Schrag SJ, Arvay M, Humphrys M, Ravel J, Adelglass J, Essink B, Musante DB, Maguire R, Gorman R, Formentini E, Mason R, Robb ML, Neuzil KM, Rapaka RR, Wolff P, Kotloff KL; SNIFF study team. Vaccine efficacy of NVX-CoV2373 against SARS-CoV-2 infection in adolescents in the USA: an ancillary study to a phase 3, observer-blinded, randomised, placebo-controlled trial. Lancet Microbe. 2025 Apr;6(4):100984. doi: 10.1016/j.lanmic.2024.100984. Epub 2025 Jan 27. PMID 39884302
- [Derived] Janes H, Fisher LH, Kee JJ, Parameswaran L, Goepfert PA, Falsey AR, Ludwig J, Magaret CA, Gilbert PB, Kublin JG, Rouphael N, Sobieszczyk ME, El Sahly HM, Baden LR, Grinsztejn B, Walsh SR, Gray GE, Kotloff KL, Gay CL, Greninger AL, Tapia MD, Hammershaimb EA, Priddy FH, Green JA, Struyf F, Dunkle L, Neuzil KM, Corey L, Huang Y. Association Between SARS-CoV-2 Viral Load and COVID-19 Vaccination in 4 Phase 3 Trials. J Infect Dis. 2024 Dec 16;230(6):1384-1389. doi: 10.1093/infdis/jiae400. PMID 39225478
- [Derived] Turley CB, Tables L, Fuller T, Sanders LJ, Scott H, Moodley A, Woodward Davis A, Leav B, Miller J, Schoemaker K, Vandebosch A, Sadoff J, Woo W, Cho I, Dunkle LM, Li S, van der Laan L, Gilbert PB, Follmann D, Jaynes H, Kublin JG, Baden LR, Goepfert P, Kotloff K, Gay CL, Falsey AR, El Sahly HM, Sobieszczyk ME, Huang Y, Neuzil KM, Corey L, Grinsztejn B, Gray G, Rouphael N, Luedtke A; COVID-19 Prevention Network CoVPN. Modifiers of COVID-19 vaccine efficacy: Results from four COVID-19 prevention network efficacy trials. Vaccine. 2023 Jul 25;41(33):4899-4906. doi: 10.1016/j.vaccine.2023.06.066. Epub 2023 Jun 23. PMID 37385888
- [Derived] Marchese AM, Zhou X, Kinol J, Underwood E, Woo W, McGarry A, Beyhaghi H, Anez G, Toback S, Dunkle LM. NVX-CoV2373 vaccine efficacy against hospitalization: A post hoc analysis of the PREVENT-19 phase 3, randomized, placebo-controlled trial. Vaccine. 2023 May 22;41(22):3461-3466. doi: 10.1016/j.vaccine.2023.04.054. Epub 2023 Apr 29. PMID 37127523
- [Derived] Anez G, Dunkle LM, Gay CL, Kotloff KL, Adelglass JM, Essink B, Campbell JD, Cloney-Clark S, Zhu M, Plested JS, Roychoudhury P, Greninger AL, Patel N, McGarry A, Woo W, Cho I, Glenn GM, Dubovsky F; 2019nCoV-301-Pediatric Expansion Study Group. Safety, Immunogenicity, and Efficacy of the NVX-CoV2373 COVID-19 Vaccine in Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e239135. doi: 10.1001/jamanetworkopen.2023.9135. PMID 37099299
- [Derived] Anez G, Dunkle LM, Gay CL, Kotloff KL, Adelglass JM, Essink B, Campbell JD, Cloney-Clark S, Zhu M, Plested JS, Roychoudhury P, Greninger AL, Patel N, McGarry A, Woo W, Cho I, Glenn GM, Dubovsky F; 2019nCoV-301 - Pediatric Expansion Study Group. Safety, Immunogenicity and Efficacy of NVX-CoV2373 in Adolescents in PREVENT-19: A Randomized, Phase 3 Trial. medRxiv [Preprint]. 2022 Sep 21:2022.09.20.22279903. doi: 10.1101/2022.09.20.22279903. PMID 36172135
- [Derived] Dunkle LM, Kotloff KL, Gay CL, Anez G, Adelglass JM, Barrat Hernandez AQ, Harper WL, Duncanson DM, McArthur MA, Florescu DF, McClelland RS, Garcia-Fragoso V, Riesenberg RA, Musante DB, Fried DL, Safirstein BE, McKenzie M, Jeanfreau RJ, Kingsley JK, Henderson JA, Lane DC, Ruiz-Palacios GM, Corey L, Neuzil KM, Coombs RW, Greninger AL, Hutter J, Ake JA, Smith K, Woo W, Cho I, Glenn GM, Dubovsky F; 2019nCoV-301 Study Group. Efficacy and Safety of NVX-CoV2373 in Adults in the United States and Mexico. N Engl J Med. 2022 Feb 10;386(6):531-543. doi: 10.1056/NEJMoa2116185. Epub 2021 Dec 15. PMID 34910859